CLINICAL TRIAL: NCT05390996
Title: Implant Stability Changes In Dental Implants Installed By Osseodensification and Conventional Methods: A Randomized Controlled Study
Brief Title: Implant Stability Changes In Dental Implants Installed By Osseodensification and Conventional Methods
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Noor Abdulhakeem, Msc.student, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: dental implant
Record Dates: First submitted 2022-05-07; First posted 2022-05-25 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Dental Implant Stability

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- condensation drilling technique (Active Comparator): condensation of bone (osseodensefecation technique)
  Interventions: Other: dental implant placement
- conventional drilling technique (Sham Comparator): control group
  Interventions: Other: dental implant placement

INTERVENTIONS:
Other: dental implant placement — dental implant placement by using a different drilling techniques

SUMMARY:
The aim of this study is to evaluate the effect of Osseodensification on implant stability during the healing period The objective of this study is to compare between dental implant stability after osteotomy site preparation using osseodensification technique and conventional drilling technique immediately after implant installation (primary stability) , 6 week after the insertion of implant and 12 weeks later (secondary stability)

ELIGIBILITY:
Inclusion Criteria:

1. medically fit patients ≥ 18 years of age including both genders
2. alveolar ridges of sufficient vertical and horizontal dimensions
3. bone density less than 850 Hounsfield units (HU) which corresponds to D3-D5 bone density according to Misch bone classification based on preoperative CBCT findings

Exclusion Criteria:

1. Patients with high bone density (more than 850 HU which corresponds to D1 and D2 according to Misch classification are not suitable for osseodensification.
2. Patient with severe buccal plate undercut or concavity
3. Active infection or inflammation in the implant zone
4. Presence of any uncontrolled systemic diseases.
5. Any patient need advance treatment such as sinus lifting and bone augmentation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2022-01-05 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
primary stability | 0 day (baseline)
  Mean implant stability between different comparators following implants insertion by using resonance frequency analysis scaled from 1 to 100
stability at the dip period | 6 week post surgery
  Mean implant stability between different comparators following implants insertion by using resonance frequency analysis scaled from 1 to 100
secondary stability | 12 week post surgery
  Mean implant stability between different comparators following implants insertion by using resonance frequency analysis scaled from 1 to 100

CONTACTS AND LOCATIONS:
Overall Officials: Salwan Y Bede, BDS,FIMBS, Principal Investigator — University of Bagh
Locations (1):
- Baghdad University, Baghdad, Babalmatham, Iraq